CLINICAL TRIAL: NCT06045494
Title: A Randomized, Open-Label Trial of the Efficacy of Treatment for Helicobacter Pylori Infection in Preschooler by Yoghurt With LG21
Brief Title: The Efficacy of Treatment for Helicobacter Pylori Infection in Preschooler by Yoghurt With LG21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meiji China Investment Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-SM-04-MJ-001
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: H. Pylori Infection
Keywords: Meiji Yoghurt LG21; Helicobacter pylori stool antigen test; Preschooler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meiji Yogurt Group (Active Comparator): Meiji LG21 yogurt: 180 g/bottle, main ingredients:
  Raw milk, water, sugar, skim milk powder, food additives (hydroxypropyl distarch phosphate, pectin), cream, whey protein powder, food flavor, Lactobacillus grigi, Lactobacillus bulgaricus, Streptococcus thermophilus.
  Interventions: Dietary Supplement: Meiji Yogurt Group
- Blank Control Group (No Intervention): No interventional product for this arm

INTERVENTIONS:
Dietary Supplement: Meiji Yogurt Group — Participants in this arm need to eat assigned product for 12 weeks, one bottle each day.
  Arms: Meiji Yogurt Group

SUMMARY:
The goal of this randomized, open-label, interventional trial is to study the efficacy of treatment for Helicobacter Pylori Infection in Preschooler aged 4-6 by Meiji Yoghurt with LG21. The main question it aims to answer is:

- whether the treatment by Meiji Yoghurt LG21 is effective by stool antigen (HpSA) test

140 qualified participants will be enrolled and randomized into 2 groups of the same size (product study group and blank control group). Participants of the product study group will need to eat assigned Meiji Yoghurt for 12 weeks, one bottle each day, while participants of the blank control group won't receive any intervention during the study. Four visits will be made for all participants, and relevant clinical data will be captured and recorded into CTMS (Clinical Trial Management System) for statistical analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Preschooler aged 4-6 years
* H. pylori positive
* Drink milk or milk beverages regularly (more than three times a week) before joining the study
* ICF signed
* Parents or guardians agree not to participate in other interventional clinical studies during this study

Exclusion Criteria:

* Has potential metabolic class or chronic disease
* Use of antibiotics within 7 days before randomization (as judged by the trial responsible physician)
* People who have been treated for eradication of Helicobacter pylori
* Pharmaceuticals, medicinal skin care products (medical external products) and health foods that may affect gastric symptoms have been commonly used since more than one month ago
* Already under digestive system treatment
* Has lactose intolerance or protein allergy
* Those whose families had plans to leave Jinhua City during the study period
* Fails to comply with the provisions of the protocol
* Those who are deemed unsuitable as subjects by the physician

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
H. pylori-negative conversion rate and the levels of H. pylori antigen measured and confirmed through fecal H. pylori antigen tests at each visit. | baseline day 0, day 42, day 84, day 112
  The stool of the participants will be assessed by Helicobacter pylori Stool Antigen Test (HpSA) on baseline day 0, day 42, day 84, and day 112. A negative result indicates that participant is infection-free.

SECONDARY OUTCOMES:
Gastrointestinal symptom scores | baseline day 0, day 42, day 84, day 112
  A questionnaire will be administered in which parents will report on 12 gastrointestinal symptoms related to their child's esophagus, stomach, and lower abdomen over the past week on baseline day 0, day 42, day 84, and day 112. The following symptoms will be evaluated using a 7-point Likert scale
Stool frequency score (using the Bristol stool scale) | baseline day 0, day 42, day 84, day 112
  A questionnaire will be administered in which parents will report their child's stool frequency over the past week on baseline day 0, day 42, day 84, and day 112. Stool frequency will be assessed using a 5-point Likert scale.
Stool consistency (using the Bristol stool scale) | baseline day 0, day 42, day 84, day 112
  A questionnaire will be administered in which parents will report their child's stool consistency over the past week on baseline day 0, day 42, day 84, and day 112. The stool of the participants will be assessed by Bristol Stool Scale, type 1 to type 7, mapping to a score from 1 to 7.
The problem behavior scores (using the Child Behavior Checklist, CBCL) | baseline day 0, day 84
  The Chinese version of the Preschool Child Behavior Checklist (CBCL) (1.5-5) will be used on baseline day 0 and day 84. The parents will be asked to describe their child's behavior now or within the past 2 months on a Likert scale.
Salivary amylase and cortisol levels | baseline day 0, day 84
  The concentrations of salivary cortisol (µg/L) and salivary amylase (µM/L)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhuang, MD, Principal Investigator — Jinhua Wenrong Hospital; Toshihiro Otsu, PhD, Principal Investigator — Meiji China Investment Co.,Ltd
Locations (1):
- Kaitai Biotech Lab, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding SZ, Du YQ, Lu H, Wang WH, Cheng H, Chen SY, Chen MH, Chen WC, Chen Y, Fang JY, Gao HJ, Guo MZ, Han Y, Hou XH, Hu FL, Jiang B, Jiang HX, Lan CH, Li JN, Li Y, Li YQ, Liu J, Li YM, Lyu B, Lu YY, Miao YL, Nie YZ, Qian JM, Sheng JQ, Tang CW, Wang F, Wang HH, Wang JB, Wang JT, Wang JP, Wang XH, Wu KC, Xia XZ, Xie WF, Xie Y, Xu JM, Yang CQ, Yang GB, Yuan Y, Zeng ZR, Zhang BY, Zhang GY, Zhang GX, Zhang JZ, Zhang ZY, Zheng PY, Zhu Y, Zuo XL, Zhou LY, Lyu NH, Yang YS, Li ZS; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology, and Chinese Alliance for Helicobacter pylori Study. Chinese Consensus Report on Family-Based Helicobacter pylori Infection Control and Management (2021 Edition). Gut. 2022 Feb;71(2):238-253. doi: 10.1136/gutjnl-2021-325630. Epub 2021 Nov 26. PMID 34836916
- [Background] Liu WZ, Xie Y, Lu H, Cheng H, Zeng ZR, Zhou LY, Chen Y, Wang JB, Du YQ, Lu NH; Chinese Society of Gastroenterology, Chinese Study Group on Helicobacter pylori and Peptic Ulcer. Fifth Chinese National Consensus Report on the management of Helicobacter pylori infection. Helicobacter. 2018 Apr;23(2):e12475. doi: 10.1111/hel.12475. Epub 2018 Mar 7. PMID 29512258
- [Background] Cheng ZY, Gao Y, Mao F, Lin H, Jiang YY, Xu TL, Sun C, Xin L, Li ZS, Wan R, Zhou MG, Wang LW; China Gastrointestinal Health Expert Group (CGHEG). Construction and results of a comprehensive index for gastrointestinal health monitoring in China: a nationwide study. Lancet Reg Health West Pac. 2023 Jun 29;38:100810. doi: 10.1016/j.lanwpc.2023.100810. eCollection 2023 Sep. PMID 37435093
- [Background] Boonyaritichaikij S, Kuwabara K, Nagano J, Kobayashi K, Koga Y. Long-term administration of probiotics to asymptomatic pre-school children for either the eradication or the prevention of Helicobacter pylori infection. Helicobacter. 2009 Jun;14(3):202-7. doi: 10.1111/j.1523-5378.2009.00675.x. PMID 19702850